CLINICAL TRIAL: NCT03638414
Title: ePainQ - a Web-based Pain Self-management System for Patients Undergoing Surgery for Breast Cancer: Feasibility Study
Brief Title: ePainQ - Feasibility Study
Acronym: ePainQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS18/107321
Record Dates: First submitted 2018-06-04; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Interventional Treatment (Experimental): This group will be given the ePainQ questionnaire and an interview.
  Interventions: Other: ePainQ questionnaire
- Group 2 - Usual care (No Intervention): This group will be receiving normal routine care without the study intervention

INTERVENTIONS:
Other: ePainQ questionnaire — This is a questionnaire which will be given to the intervention group about their perceptions of treatment. It will be online.
  Arms: Group 1 - Interventional Treatment

SUMMARY:
This is a feasibility study of a web-based pain self-management system aimed at providing support for acute postoperative pain and enhancing patient care. The ePainQ symptom questionnaire provides patients with immediate graded advice dependent on severity of issues reported. Information about self-managing these issues are provided via instructions in ePainQ with hyperlinks to more detailed advice on the ePainQ website. Patients log on daily postoperatively to complete the symptom questionnaire.

Women with invasive/non-invasive breast carcinoma due to be treated by surgery with curative intent will be approached to take part in this study. We will invite consecutive eligible patients, consenting as many willing patients as possible within a fixed 12 month recruitment period. There are 2 arms to the study: intervention -using ePainQ intervention & standard care and a cohort (control) arm, which will be standard care only.

Primary aim: To test the feasibility of a web-based pain self-management system for breast cancer patients undergoing surgery Secondary aims: 1. a) Examine preliminary effectiveness of the system (impact on outcome measures, pain etc.) b) Explore the potential associations between breast density, post-surgical scarring and pain and outcomes 2. To explore staff use and perceived usefulness of ePainQ in clinical consultations.

ELIGIBILITY:
Inclusion Criteria:

Aged over 18 years of age at the time of diagnosis of cancer Primary operable (TNM categories: T1, T2, T3, N0, N1, M0; invasive breast cancer or non-invasive breast cancer (diagnosed on core biopsy or diagnostic incision biopsy) Ability to give informed consent Access to the internet (those without access to the internet may participate in the cohort arm) Ability to speak and write english

Exclusion Criteria:

* Male Disease unsuitable for surgery e.g. inoperable, locally recurrent or metastatic disease Previously treated invasive breast cancer There will be a restriction to people who are able to speak/read English. This is due to lack of funding for translation of study documents Pregnant women Patients without capacity to consent or those with a major psychiatric disorder No internet access (those without access to the internet may participate in the cohort arm)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female patients are eligible as this is only run in the female breast clinic.
Enrollment: 25 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Successful completion of the ePainQ questionnaire | 10 months from initial completion of questionnaire to feedback about experience
  Feasibility of the ePainQ system is the primary outcome measure for the study. This will be examined in terms of:
  1. Patient uptake rates
  2. Patient engagement with/use of the system (e.g. log ins and completed questionnaires)
  3. Patient retention rates
  4. Representativeness of the participants (clinically and sociodemographic)
  5. Patient feedback on perceived usability via qualitative interviews
  6. System 'running burden' for the provider

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No